CLINICAL TRIAL: NCT02377583
Title: Hypothalamo-pituitary Adrenal Axis Activity: Relation With Neuropsychological Consequences in Type 1 Diabetes in Childhood. The CORTICODIAB Study
Brief Title: Hypothalamo-pituitary Adrenal Axis Activity and Neuropsychological Consequences in Type 1 Diabetes in Childhood
Acronym: CORTICODIAB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2011/24
Record Dates: First submitted 2015-02-25; First posted 2015-03-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 20ml blood sample in order to evaluate:
  * NR3C1 (GR) gene
  * NR3C2 (MR) gene
  * FKBP5 gene
  * CRH gene
  * CRHR1 gene
  * CBG gene
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Diabetic children: * physical examination
  * Glucocorticoid sensitivity index
  * DNA sample
  * Anxiety and depression questionnaires
  * depression questionnaire
  * MRI
- Controls: * physical examination
  * Glucocorticoid sensitivity index
  * DNA sample
  * Anxiety and depression questionnaires
  * depression questionnaire
  * MRI
  * Laboratory tests

SUMMARY:
The general objective is to precise the role of HPA axis activity in neuropsychological consequences of type 1 diabetes. The investigators hypothesize that hyperactivity of HPA axis is associated with higher scores of depression and changes in hippocampal volume and mean diffusion.

DETAILED DESCRIPTION:
* Background: Type 1 diabetes could be associated with hyperactivity of hypothalamo-pituitary adrenal (HPA) axis. Type 1 diabetes is associated with higher frequency neuropsychological consequences as mood disorders and structural changes in brain, particularly in hippocampus.
* Purpose: To describe the association between HPA axis activity and anxiety and depression scores in 6-12 year's old diabetes children.
* Abstract: The general objective is to precise the role of HPA axis activity in neuropsychological consequences of type 1 diabetes. The investigators hypothesize that hyperactivity of HPA axis is associated with higher scores of depression and changes in hippocampal volume and mean diffusion.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic group:

  * diabetes for 1 year
  * 6-12 year's old
  * included in ISIS-DIAB protocol.
* Control group:

  * brother or sister of a diabetic children
  * 6-12 year's old.

Exclusion Criteria:

* Per os or inhaled corticoid in the previous month of inclusion.
* Acute infectious disease in the previous week of inclusion.
* Other chronic disease than diabetes type1.
* Psychiatric disorders or psychiatric treatment.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: * Age: The investigators will limit the study to children at least 6 years, to ensure the successful completion of saliva samples and MRI without anesthesia. The investigators limit themselves to prepubescent children do not have to take into account the influence of sex steroids on the AC activity.
  * Gender: Although it is expected differences in hippocampal volume and CA activity between boys and girls, the relationship between these two variables is not necessarily different for boys and girls. Thus, the inclusion of both sexes in the analysis is not necessarily problematic, and will be more informative. So it has been finally decided to include boys and girls in the sample of subjects undergoing MRI.
  * Population control: The constitution of a control group from the siblings will enable to study the specific effect of diabetes on anxiety and depression, regardless of the children's education mode in the same family environment.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2012-08; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Mean of nocturnal urinary free cortisol during 5 days. | During 5 days after the inclusion
Depression (CDI) score | At the inclusion

SECONDARY OUTCOMES:
Mean of awakening salivary cortisol and mean of nocturnal urinary cortisol metabolites during 5 days | During 5 days after the inclusion
Profiles of glucocorticoid sensitive genes expressed in peripheral blood mononuclear cells. | At the inclusion
Anxiety (STAI) score | At the inclusion
Polymorphisms of genes involved in HPA axis activity | At the inclusion
Hippocampal volume and mean diffusion | At the inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Paul PEREZ, Doctor, Study Chair — University Hospital, Bordeaux
Locations (3):
- France (3):
  - Service d'endocrinologie pédiatrique CHG Bayonne Centre Hospitalier de la Côte Basque, Bayonne, Aquitaine
  - CHU de Bordeaux Hôpital Pellegrin, Bordeaux, Aquitaine
  - Service d'endocrinologie pédiatrique - Hôpital de la mère et de l'enfant - CHU de LIMOGES, Limoges, Limousin